CLINICAL TRIAL: NCT05439967
Title: Investigation of The Effects of Augmented and Virtual Reality Gait Training on Balance and Walking in Patients With Parkinson's Disease
Brief Title: The Effects of Augmented and Virtual Reality Gait Training on Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fettah Saygılı, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-PD C-Mill
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Exercise; Virtual Reality; Balance; Gait
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Augmented and Virtual Reality Gait and balanceTraining
- Conventional Training (Active Comparator)
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Augmented and Virtual Reality Gait and balanceTraining — C-Mill VR+ device used for training. The training was carried out 3 days a week for 6 weeks, with each exercise session lasting approximately 1.5 hours, accompanied by a physiotherapist. Training started with conventional exercises, continued with C-Mill VR+ training, and ended with stretching and relaxation exercises. The patients in the intervention group were applied the exercises with the same principles with conventional training, except the exercises performed in standing and walking. Patients performed 10 exercises in AR and VR gait training for 4 minutes and resting the individuals by sitting for 1 minute between exercises.
  Arms: Intervention
Other: Conventional Training — Conventional training was applied to the patients in the control group. Conventional training was planned taking into account the following goals: increasing mobility by improving the impaired kinesthetic sensation; improving axial rotation, coordination, flexibility of soft tissues, mobility in and out of bed; increasing body image perception by improving upright and proper posture; and improving balance and gait. The training was applied 3 days a week for 6 weeks, with each exercise session lasting 40-50 minutes, accompanied by a physiotherapist. Each of the exercises was done in 2 sets of 10 repetitions. In gait training, each exercise was performed for 4 minutes.
  Arms: Conventional Training

SUMMARY:
In Parkinson's Disease (PD) rehabilitation, the treadmill is used both in aerobic training and in gait training, as it provides more walking distance and can include body weight supported systems. It has been reported that the C-Mill VR+ device, which is a treadmill system with augmented and virtual reality (VR) technology, improves gait adaptation and reduces the risk of falling in individuals with early to mid-stage PD. Several publications augmented reality (AR) and VR applications in PD was focused on balance activities that do not include ambulation. In other studies in the literature, it was stated that further research are needed to better understand the effects of VR gait training on gait and balance in PD. It was also stated in these studies that the effects of VR gait training should be examined with more objective measurement methods. As a result, it is seen that there is a need for studies examining the effects of augmented and virtual reality trainings in PD with objective measurement methods. Therefore, our study aimed to examine the effects of AR and VR gait training on gait and balance in individuals with early to mid-stage PD.

DETAILED DESCRIPTION:
Participants included in the study will randomly divide were randomly divided into 2 groups as intervention (IG, n=15) and control (CG, n=15). IG was given augmented and virtual reality gait training together with conventional training (CT). CG was given CT only. The training was applied 3 days per week for 6 weeks in both groups. All evaluations will be made by the same physiotherapist by meeting with participants face to face. Inclusion in the research will be on a voluntary basis. As outcome measures, motor symptoms, balance, balance confidence and gait analyses were performed before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with Parkinson's Disease by a specialist physician
* being grade 1-3 on the Hoehn and Yahr Staging Scale
* being 40 years or older; and
* individuals agreed to be included in the study after adequate information was given about the study

Exclusion Criteria:

* People who standardised Mini-Mental State Examination score < 24
* Having any cardiovascular, vestibular, musculoskeletal, or additional neurological disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS-III)-Baseline | Assessment will be conducted before intervention
  The severity of motor symptoms is evaluated with 13 items in UPDRS-III. Items are scored between 0 and 4; 0 = no impairment, 4 = severe impairment. Higher scores indicate more serious impairment
Unified Parkinson's Disease Rating Scale (UPDRS-III)-Post Intervention | Assessment will be conducted immediately after the intervention
  The severity of motor symptoms is evaluated with 13 items in UPDRS-III. Items are scored between 0 and 4; 0 = no impairment, 4 = severe impairment. Higher scores indicate more serious impairment
Hoehn and Yahr Staging Scale -Baseline | Assessment will be conducted before intervention
  H&Y defines individuals with PD in 5 different clinical stages according to their functional disability status and clinical findings. As the stage of H&Y increases, the functional disability status of patients also increases
Hoehn and Yahr Staging Scale -Post Intervention | Assessment will be conducted immediately after the intervention
  H&Y defines individuals with PD in 5 different clinical stages according to their functional disability status and clinical findings. As the stage of H&Y increases, the functional disability status of patients also increases
Huber 360° Evolution System-baseline | Assessment will be conducted before intervention
  Static and dynamic standing balance was evaluated with the Huber 360° Evolution System(LPG Systems, Valence, France), which objectively evaluated postural sway and limits of stability. Stability test and stability limit test were performed with the system. The stability test was performed by recording the amount of sway of the center of pressure (CoP) under standing on double-leg and standing on single-leg conditions. The test was performed under eyes open and eyes closed conditions. The lower values obtained as a result of the test means that the amount of sway is low and the postural stability is better. In the limits of stability test, while on standing and with fixed feet position patients are asked to shift their weight in a total of eight directions according to the trigonometric coordinate system. The high values obtained as a result of the test means that the amount of CoP sway is high and the stability limits of the patient is good.
Huber 360° Evolution System-Post Intervention | Assessment will be conducted immediately after the intervention
  Static and dynamic standing balance was evaluated with the Huber 360° Evolution System(LPG Systems, Valence, France), which objectively evaluated postural sway and limits of stability. Stability test and stability limit test were performed with the system. The stability test was performed by recording the amount of sway of the center of pressure (CoP) under standing on double-leg and standing on single-leg conditions. The test was performed under eyes open and eyes closed conditions. The lower values obtained as a result of the test means that the amount of sway is low and the postural stability is better. In the limits of stability test, while on standing and with fixed feet position patients are asked to shift their weight in a total of eight directions according to the trigonometric coordinate system. The high values obtained as a result of the test means that the amount of CoP sway is high and the stability limits of the patient is good.
Berg Balance Scale (BBS)-Baseline | Assessment will be conducted before intervention
  Functional balance was evaluated with BBS . It consists of 14 functional activities that evaluate the static and proactive balance, in which the individual is observed directly by the evaluator in terms of desired performance. Each item is scored between 0 (inability to perform the activity) and 4 (doing the activity completely independently) according to the performance of the individual to perform the desired functional activity according to the time and distance conditions of the test. BBS is scored between 0 and 56, and higher test scores mean that the individual's balance is better
Berg Balance Scale-Post Intervention | Assessment will be conducted immediately after the intervention
  Functional balance was evaluated with BBS . It consists of 14 functional activities that evaluate the static and proactive balance, in which the individual is observed directly by the evaluator in terms of desired performance. Each item is scored between 0 (inability to perform the activity) and 4 (doing the activity completely independently) according to the performance of the individual to perform the desired functional activity according to the time and distance conditions of the test. BBS is scored between 0 and 56, and higher test scores mean that the individual's balance is better
Activities-specific Balance Confidence Scale (ABC) -Baseline | Assessment will be conducted before intervention
  The level of confidence that an individual feels during activities of daily living related to balance was evaluated with ABC. With 16 questions asked directly to the individual by the evaluator, the level of confidence ranged from 0% (totally unsafe) to 100% (totally safe). The total score is determined by summing the values of 16 items and dividing by 16, which is the total number of question items. A total score between 0 and 49 indicates a low functional level, between 50 and 80 indicates a moderate functional level, and between 81 and 100 indicates a high functional level.
Activities-specific Balance Confidence Scale (ABC) -Post Intervention | Assessment will be conducted immediately after the intervention
  The level of confidence that an individual feels during activities of daily living related to balance was evaluated with ABC. With 16 questions asked directly to the individual by the evaluator, the level of confidence ranged from 0% (totally unsafe) to 100% (totally safe). The total score is determined by summing the values of 16 items and dividing by 16, which is the total number of question items. A total score between 0 and 49 indicates a low functional level, between 50 and 80 indicates a moderate functional level, and between 81 and 100 indicates a high functional level.
Spatio-temporal gait analysis -Baseline | Assessment will be conducted before intervention
  In the evaluation of spatio-temporal parameters of gait, patients were asked to walk on the platform of the C-Mill VR+ device for 3 minutes at the highest confident speed they felt safe. Right-left step lengths, stride length, and step width were recorded in meters from the spatial parameters, while the right-left stance phase duration, right-left swing phase duration and total double support phase duration were recorded in seconds for the evaluation of temporal parameters. Additionally, walking speed and distance were recorded during these analyses.
Spatio-temporal gait analysis -Post Intervention | Assessment will be conducted immediately after the intervention
  In the evaluation of spatio-temporal parameters of gait, patients were asked to walk on the platform of the C-Mill VR+ device for 3 minutes at the highest confident speed they felt safe. Right-left step lengths, stride length, and step width were recorded in meters from the spatial parameters, while the right-left stance phase duration, right-left swing phase duration and total double support phase duration were recorded in seconds for the evaluation of temporal parameters. Additionally, walking speed and distance were recorded during these analyses.
Timed Up and Go Test (TUG)- Baseline | Assessment will be conducted before intervention
  Functional mobility was assessed with TUG. The patient was asked to stand up from the chair with the "walk" command, walk 3 m, turn around and sit back on the chair. The test was carried out on a flat 3 meter surface. In addition, TUG has been shown to be highly reliable in PD.
Timed Up and Go Test (TUG)- Post Intervention | Assessment will be conducted immediately after the intervention
  Functional mobility was assessed with TUG. The patient was asked to stand up from the chair with the "walk" command, walk 3 m, turn around and sit back on the chair. The test was carried out on a flat 3 meter surface. In addition, TUG has been shown to be highly reliable in PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No